CLINICAL TRIAL: NCT05430698
Title: PD-1 Antibody Plus Gemcitabine and Oxaliplatin (GEMOX) as Postoperative Adjuvant Therapy in Perihilar Cholangiocarcinoma Patients With Positively Metastatic Lymph Nodes : a Single Arm, Phase II Trial
Brief Title: PD-1 Antibody Plus GEMOX as Postoperative Adjuvant Therapy in Perihilar Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LX-GY-2022010
Record Dates: First submitted 2022-05-29; First posted 2022-06-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-07

CONDITIONS: Perihilar Cholangiocarcinoma
Keywords: PD-1; GEMOX; Perihilar Cholangiocarcinoma; Positively Metastatic Lymph Nodes
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PD-1antibody plus GEMOX (Experimental): PD-1 antibody plus GEMOX was given as postoperative adjuvant therapy
  Interventions: Drug: PD-1antibody plus GEMOX

INTERVENTIONS:
Drug: PD-1antibody plus GEMOX — 1. PD-1 antibody，200mg，D1，intravenous infusion, the administration time is 60 (+15) minutes.
  2. GEMOX chemotherapy : gemcitabine 1000mg/m2,D1，D8；oxaliplatin 100mg/m2,D1，intravenous infusion.
  3. Three weeks is a course of treatment,a total of 6-8 courses.

SUMMARY:
This is an open-label,single center,non-randomized,single arm exploratory study. The objective of this study is to evaluate the efficacy and safety of PD-1 antibody plus GEMOX as postoperative adjuvant therapy in perihilar cholangiocarcinoma with positively metastatic lymph nodes.

DETAILED DESCRIPTION:
For perihilar cholangiocarcinoma, radical surgical treatment, such as major hepatectomy combined with total caudate lobe and extrahepatic bile duct resection, remain the potential modality for cure. However, the lymph node tumor metastasis is an independent risk factor for prognosis after radical resection for this disease without distant metastasis. As reported by Nagoya University, Japan, the patients without lymph node tumor metastasis, the 5-year survival rate could reach as high as 67.1% after R0 resection, but the 5-year survival rate was only 22.1% for the patients with lymph node tumor metastasis after R0 resection. Thus, it is urgent to look for an effective adjuvant therapy treatment for these patients with lymph node tumor metastasis. Fluoropyrimidine-based or gemcitabine-based chemotherapy was recommended for these patients by NCCN guidelines. Studies have shown that Gemox chemotherapy (oxaliplatin + gemcitabine) in patients with resected biliary tract cancer has a good benefit in overall survival. However, for extrahepatic cholangiocarcinoma with lymph nodes metastasis, the benefit was limited. In recent years, immunotherapy, such as PD-1 or PD-L1 monoclonal antibody, combined with chemotherapy have shown better results in the palliative treatment of un-resectable biliary tract tumor. However, there is no report on combined immunotherapy with chemotherapy as adjuvant therapy in perihilar cholangiocarcinoma with lymph node tumor metastasis after R0 resection.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must sign an informed consent form;
2. Age 18-75 years old, both male and female;
3. ECOG performance status score (PS score) 0 or 1 point;
4. Child-Pugh score A period;
5. Perihepatic cholangiocarcinoma with negative margins and positively metastatic lymph nodes confirmed by histopathology. Abdominal positively metastatic lymph nodes region is not limited. The 16 groups of microscopically positively metastatic lymph nodes can be included.
6. Have not received any systemic treatment within 6 months;
7. The functional indicators of important organs meet the following requirements (1)Neutrophils≥1.5*109/L; platelets≥100*109/L; hemoglobin≥9g/dl; serum albumin≥3g/dl; (2)Thyroid-stimulating hormone (TSH) ≤ 2 times the upper limit of normal, and T3 and T4 are in the normal range; (3)Bilirubin ≤ 1.5 times the upper limit of normal; ALT and AST ≤ 3 times the upper limit of normal; (4)Serum creatinine ≤ 1.5 times the upper limit of normal, and creatinine clearance ≥ 60ml/min (calculated by Cockcroft-Gault formula); 8. The subject has at least 1 measurable lesion (according to RECIST1.1);
8. For women who are not breastfeeding or pregnant, use contraception during treatment or 12 months after the end of treatment.

Exclusion Criteria:

1. Unresectable PHC patients or postoperative diagnosis of PHC recurrence and metastasis ;
2. Past or simultaneous suffering from other malignant tumors, except for fully treated non-melanoma skin cancer, cervical carcinoma in situ, and thyroid papillary carcinoma;
3. Have used gemcitabine-based chemotherapy or have used PD-1 monoclonal antibody or PD-L1 monoclonal antibody treatment within 6 months;
4. Severe cardiopulmonary and renal dysfunction;
5. Hypertension that is difficult to control with drugs (systolic blood pressure (BP) ≥140 mmHg and/or diastolic blood pressure ≥90mmHg) (based on the average of ≥3 BP readings obtained by ≥2 measurements);
6. Abnormal coagulation function (PT>14s), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy;
7. After antiviral treatment, HBV DNA>2000 copies/ml, HCV RNA>1000;
8. A history of esophageal and gastric varices, significant clinically significant bleeding symptoms or a clear tendency to appear within 3 months before enrollment;
9. Active infections requiring systemic treatment; patients with active tuberculosis infection within 1 year before enrollment; a history of active tuberculosis infection more than 1 year before enrollment, and no formal anti-tuberculosis treatment or tuberculosis Still in the active period;
10. Human immunodeficiency virus (HIV, HIV1/2 antibody) positive;
11. A history of psychotropic drug abuse, alcohol or drug abuse;
12. Known to have a history of severe allergies to any monoclonal antibodies, platinum drugs, or gemcitabine;
13. Other factors judged by the investigator may affect the safety of the subjects or the compliance of the trial. Such as serious diseases (including mental illness) that require combined treatment, serious laboratory abnormalities, or other family or social factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The 12-month relapse-free survival rate | 12 months
  Relapse-free survival rate in perihilar cholangiocarcinoma with positively metastatic lymph nodes.

SECONDARY OUTCOMES:
The 12-month overall survival rate | 12 months
  Overall survival rate in perihilar cholangiocarcinoma with positively metastatic lymph nodes.
The 60-month overall survival rate | 60 months
  Overall survival rate in perihilar cholangiocarcinoma with positively metastatic lymph nodes.
Relapse-free survival | 60 months
  RFS is defined as the time from resection to relapse or death from any cause, whichever occurred first.
Overall survival | 60 months
  OS is defined as the time from resection to death from any cause.
Percentage of participants with adverse events (AEs) | 12 months
  Number of participants who experienced an adverse event (AE)

CONTACTS AND LOCATIONS:
Overall Officials: Chao Liu, PhD, Principal Investigator — Department of Biliary and Pancreatic Surgery, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeOliveira ML, Cunningham SC, Cameron JL, Kamangar F, Winter JM, Lillemoe KD, Choti MA, Yeo CJ, Schulick RD. Cholangiocarcinoma: thirty-one-year experience with 564 patients at a single institution. Ann Surg. 2007 May;245(5):755-62. doi: 10.1097/01.sla.0000251366.62632.d3. PMID 17457168
- [Background] Kang MJ, Lee JL, Kim TW, Lee SS, Ahn S, Park DH, Lee SS, Seo DW, Lee SK, Kim MH. Randomized phase II trial of S-1 and cisplatin versus gemcitabine and cisplatin in patients with advanced biliary tract adenocarcinoma. Acta Oncol. 2012 Sep;51(7):860-6. doi: 10.3109/0284186X.2012.682628. Epub 2012 May 6. PMID 22559158
- [Background] Groot Koerkamp B, Wiggers JK, Allen PJ, Besselink MG, Blumgart LH, Busch OR, Coelen RJ, D'Angelica MI, DeMatteo RP, Gouma DJ, Kingham TP, Jarnagin WR, van Gulik TM. Recurrence Rate and Pattern of Perihilar Cholangiocarcinoma after Curative Intent Resection. J Am Coll Surg. 2015 Dec;221(6):1041-9. doi: 10.1016/j.jamcollsurg.2015.09.005. Epub 2015 Sep 15. PMID 26454735
- [Background] Abdel-Rahman O, Elsayed Z, Elhalawani H. Gemcitabine-based chemotherapy for advanced biliary tract carcinomas. Cochrane Database Syst Rev. 2018 Apr 6;4(4):CD011746. doi: 10.1002/14651858.CD011746.pub2. PMID 29624208
- [Background] Ebata T, Hirano S, Konishi M, Uesaka K, Tsuchiya Y, Ohtsuka M, Kaneoka Y, Yamamoto M, Ambo Y, Shimizu Y, Ozawa F, Fukutomi A, Ando M, Nimura Y, Nagino M; Bile Duct Cancer Adjuvant Trial (BCAT) Study Group. Randomized clinical trial of adjuvant gemcitabine chemotherapy versus observation in resected bile duct cancer. Br J Surg. 2018 Feb;105(3):192-202. doi: 10.1002/bjs.10776. PMID 29405274
- [Background] Nassour I, Mokdad AA, Porembka MR, Choti MA, Polanco PM, Mansour JC, Minter RM, Wang SC, Yopp AC. Adjuvant Therapy Is Associated With Improved Survival in Resected Perihilar Cholangiocarcinoma: A Propensity Matched Study. Ann Surg Oncol. 2018 May;25(5):1193-1201. doi: 10.1245/s10434-018-6388-7. Epub 2018 Feb 27. PMID 29488187
- [Background] Edeline J, Benabdelghani M, Bertaut A, Watelet J, Hammel P, Joly JP, Boudjema K, Fartoux L, Bouhier-Leporrier K, Jouve JL, Faroux R, Guerin-Meyer V, Kurtz JE, Assenat E, Seitz JF, Baumgaertner I, Tougeron D, de la Fouchardiere C, Lombard-Bohas C, Boucher E, Stanbury T, Louvet C, Malka D, Phelip JM. Gemcitabine and Oxaliplatin Chemotherapy or Surveillance in Resected Biliary Tract Cancer (PRODIGE 12-ACCORD 18-UNICANCER GI): A Randomized Phase III Study. J Clin Oncol. 2019 Mar 10;37(8):658-667. doi: 10.1200/JCO.18.00050. Epub 2019 Feb 1. PMID 30707660
- [Background] Primrose JN, Fox RP, Palmer DH, Malik HZ, Prasad R, Mirza D, Anthony A, Corrie P, Falk S, Finch-Jones M, Wasan H, Ross P, Wall L, Wadsley J, Evans JTR, Stocken D, Praseedom R, Ma YT, Davidson B, Neoptolemos JP, Iveson T, Raftery J, Zhu S, Cunningham D, Garden OJ, Stubbs C, Valle JW, Bridgewater J; BILCAP study group. Capecitabine compared with observation in resected biliary tract cancer (BILCAP): a randomised, controlled, multicentre, phase 3 study. Lancet Oncol. 2019 May;20(5):663-673. doi: 10.1016/S1470-2045(18)30915-X. Epub 2019 Mar 25. PMID 30922733
- [Background] Ueno M, Ikeda M, Morizane C, Kobayashi S, Ohno I, Kondo S, Okano N, Kimura K, Asada S, Namba Y, Okusaka T, Furuse J. Nivolumab alone or in combination with cisplatin plus gemcitabine in Japanese patients with unresectable or recurrent biliary tract cancer: a non-randomised, multicentre, open-label, phase 1 study. Lancet Gastroenterol Hepatol. 2019 Aug;4(8):611-621. doi: 10.1016/S2468-1253(19)30086-X. Epub 2019 May 17. PMID 31109808
- [Background] Banales JM, Marin JJG, Lamarca A, Rodrigues PM, Khan SA, Roberts LR, Cardinale V, Carpino G, Andersen JB, Braconi C, Calvisi DF, Perugorria MJ, Fabris L, Boulter L, Macias RIR, Gaudio E, Alvaro D, Gradilone SA, Strazzabosco M, Marzioni M, Coulouarn C, Fouassier L, Raggi C, Invernizzi P, Mertens JC, Moncsek A, Ilyas SI, Heimbach J, Koerkamp BG, Bruix J, Forner A, Bridgewater J, Valle JW, Gores GJ. Cholangiocarcinoma 2020: the next horizon in mechanisms and management. Nat Rev Gastroenterol Hepatol. 2020 Sep;17(9):557-588. doi: 10.1038/s41575-020-0310-z. Epub 2020 Jun 30. PMID 32606456
- [Background] Chen X, Wu X, Wu H, Gu Y, Shao Y, Shao Q, Zhu F, Li X, Qian X, Hu J, Zhao F, Mao W, Sun J, Wang J, Han G, Li C, Xia Y, Seesaha PK, Zhu D, Li H, Zhang J, Wang G, Wang X, Li X, Shu Y. Camrelizumab plus gemcitabine and oxaliplatin (GEMOX) in patients with advanced biliary tract cancer: a single-arm, open-label, phase II trial. J Immunother Cancer. 2020 Nov;8(2):e001240. doi: 10.1136/jitc-2020-001240. PMID 33172881
- [Background] Itano O, Takemura Y, Kishida N, Tamagawa E, Shinozaki H, Ikeda K, Urakami H, Ei S, Hayatsu S, Suzuki K, Sakuragawa T, Ishii M, Shito M, Aiura K, Fujisaki H, Takano K, Matsui J, Minagawa T, Shinoda M, Kitago M, Abe Y, Yagi H, Oshima G, Hori S, Kitagawa Y. A prospective feasibility study of one-year administration of adjuvant S-1 therapy for resected biliary tract cancer in a multi-institutional trial (Tokyo Study Group for Biliary Cancer: TOSBIC01). BMC Cancer. 2020 Jul 23;20(1):688. doi: 10.1186/s12885-020-07185-6. PMID 32703191
- [Background] Nakahashi K, Ebata T, Yokoyama Y, Igami T, Mizuno T, Yamaguchi J, Onoe S, Watanabe N, Nagino M. How long should follow-up be continued after R0 resection of perihilar cholangiocarcinoma? Surgery. 2020 Oct;168(4):617-624. doi: 10.1016/j.surg.2020.04.068. Epub 2020 Jul 19. PMID 32665142
- [Background] Gao H, Tian T, Li S, Zhang Y, Fu X, Zheng X, Liu N, Jiang A, Ren M, Zhang X, Liang X, Ruan Z, Geng Z, Yao Y. Efficacy Analysis of Adjuvant Chemotherapy with Gemcitabine Plus Platinum or S-1 in Biliary Tract Carcinoma: A Multi-Center Retrospective Study. Cancer Manag Res. 2021 Jan 29;13:889-898. doi: 10.2147/CMAR.S290083. eCollection 2021. PMID 33542660